CLINICAL TRIAL: NCT02332681
Title: Osteoporosis and Knee Insufficiency Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Sponsor
Other Study IDs: 38151514.8.0000.5404
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporosis; Osteoporotic Fractures; Osteonecrosis
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- With insufficiency fracture: Patients with acute pain that sustained a knee insufficiency fracture
- Without insufficiency fracture: Patients with acute pain that did not sustained a knee insufficiency fracture

SUMMARY:
Osteoporosis is a systemic bone disease characterized by low bone mass and microarchitectural deterioration of bone tissue with consequent bone fragility and susceptibility to fracture. Fifty percent of women and 20% men older than 50 y.o. will have an osteoporotic fracture (fragility fracture). Fragility fracture is defined as one that results from a low-energy trauma such as a fall from body height. A previous fracture is an important predictor of a new fracture, especially in the first 5 years after initial fracture. A second fracture can be particularly devastating if it is a hip fracture. Low bone mineral density, measured by bone densitometry, as well as a previous osteoporotic fracture, are the two major risk factors for the occurrence of a new fracture.

A more rational approach currently used to minimize the costs of health care in a shorter period of time uses the strategy of firstly preventing the occurrence of secondary fracture, followed by primary prevention strategies. In this context, correct identification of fragility fractures and consequent treatment of those individuals is imperative. There are currently insufficient data about the epidemiology and evolution of other fragility fractures, also known as non-vertebral non-hip fracture (NVNH). Among these, distal radius fracture and proximal humerus fractures are the most frequent. There is a type of fracture, however, that is simply ignored by the medical community: the knee insufficiency fracture.A possible explanation for this information gap could be the fact that, until a few years ago, this entity was believed to be a osteonecrosis of the knee. Only recently it is becoming clear that the cause of pain and marrow bone edema that occur subtly in older individuals is, in fact, a insufficiency fracture. The perception that this lesion is actually a fracture is relatively new. The knee insufficiency fracture usually occurs in older individuals and those with knee osteoarthritis. This study therefore aims to evaluate whether there is a relation between knee insufficiency fracture and osteoporosis. Moreover, it is expected to find out if this fracture may be defined as a fragility fracture, electing the individuals affected by it to a prophylaxis for the occurrence of new osteoporotic fracture.

DETAILED DESCRIPTION:
Osteoporosis is a systemic bone disease characterized by low bone mass and microarchitectural deterioration of bone tissue with consequent bone fragility and susceptibility to fractures. Fifty percent of women and 20% of men older than 50 y.o. will have an osteoporotic fracture (fragility fracture). Fragility fracture is defined as one that results from a low-energy trauma such as a fall from body height. A previous fracture is an important predictor of a new fracture, especially in the first 5 years after the initial fracture. A second fracture can be particularly devastating if a hip fracture. Approximately 25% of individuals with hip fracture die in five years and only half of them recover the pre-fracture status, meaning loss of ambulation ability and independence in domestic activities. In addition, fragility fractures generate significant cost to the health system - the annual cost of osteoporotic fractures in patients older than 50 years in the United States is estimated at 1.3 billion dollar.

Low bone mineral density, measured by bone densitometry, as well as a previous osteoporotic fracture, are the two major risk factors for the occurrence of a new fracture. A crucial observation is that fracture attracts fracture, ie, individuals who had a fragility fracture are twice as likely to suffer a second fracture and half of patients with a hip fracture had previously broken another bone. Therefore, a more rational approach currently used to minimize the costs of health care more effectively and in a short time uses firstly the strategy of preventing the occurrence of secondary fracture, followed by primary prevention strategies. In this context, the correct identification of fragility fractures and the consequent treatment of individuals makes it imperative. However, it is surprising and discouraging the information that despite the huge range of currently available treatments, most patients who sustain a fragility fracture does not receive treatment.

Vertebral fractures and hip has undoubtedly the greatest impact on walking ability of the elderly, and great attention is given to these two types of fracture. Consequently, there are currently insufficient data on the epidemiology and evolution of other fragility fractures, also known as non-vertebral non-hip fracture (NVNH). Among these, distal radius and proximal humerus fractures are the most frequent. There is a type of fracture, however, that is simply ignored by the medical community: the knee insufficiency fracture. The fact that no literature study even hypothesize that this type of fracture may be a fragility fracture may be because, until a few years ago, it was believed that this entity was a osteonecrosis of the knee. The knee insufficiency fracture usually occurs in older individuals and those with knee osteoarthritis. This study therefore aims to evaluate whether a relation between the knee insufficiency fracture and osteoporosis. Moreover, it is expected to find out if this fracture may be defined as a fragility fracture, electing the individuals affected by it to a prophylaxis for the occurrence of new osteoporotic fracture.

BACKGROUND

The knee insufficiency fracture usually occurs in older individuals and those with knee osteoarthritis. Currently no literature study even suggests the hypothesis that this type of fracture may be a fragility fracture. A possible explanation for this information gap could be the fact that, until a few years ago, this entity was believed to be a osteonecrosis of the knee. Only recently it is becoming clear that the cause of pain and marrow bone edema that occur subtly in older individuals is, in fact, a insufficiency fracture. This study therefore aims to evaluate whether a relation between the knee insufficiency fracture and osteoporosis. Moreover, it is expected to find out if this fracture may be defined as a fragility fracture, electing the individuals affected by it to a prophylaxis for the occurrence of new osteoporotic fracture.

OBJECTIVES

The objective of this study is to evaluate whether there is a relationship between the knee insufficiency fracture and osteoporosis.

EXPECTED FINDINGS

Patients with knee insufficiency fracture have a higher prevalence of osteoporosis than the general population.

Patients with knee insufficiency fracture have a higher risk of having a second osteoporotic fracture

ELIGIBILITY:
Inclusion Criteria:

* patients who seek orthopedics service with sudden onset of pain in the knee;
* age of 45 y.o. or more
* acceptance by signing the informed consent form.

Exclusion Criteria:

* acute trauma of knee
* other etiologies (post-traumatic, infectious, inflammatory diseases)
* pregnant women

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients older than 45 years, with sudden joint line knee pain without high trauma history, with or without a history of osteoarthritis and / or osteoporosis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
New fracture | 12 months
  Occurrence of a new fragility fracture

SECONDARY OUTCOMES:
Bone Mineral Density | 12 months
  Evolution of bone mineral density results

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo C Campos, Phd, Principal Investigator — University of Campinas
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Result] Kanis JA, McCloskey EV, Johansson H, Cooper C, Rizzoli R, Reginster JY; Scientific Advisory Board of the European Society for Clinical and Economic Aspects of Osteoporosis and Osteoarthritis (ESCEO) and the Committee of Scientific Advisors of the International Osteoporosis Foundation (IOF). European guidance for the diagnosis and management of osteoporosis in postmenopausal women. Osteoporos Int. 2013 Jan;24(1):23-57. doi: 10.1007/s00198-012-2074-y. Epub 2012 Oct 19. PMID 23079689
- [Result] Kanis JA, Johnell O, Oden A, Sembo I, Redlund-Johnell I, Dawson A, De Laet C, Jonsson B. Long-term risk of osteoporotic fracture in Malmo. Osteoporos Int. 2000;11(8):669-74. doi: 10.1007/s001980070064. PMID 11095169
- [Result] van Staa TP, Dennison EM, Leufkens HG, Cooper C. Epidemiology of fractures in England and Wales. Bone. 2001 Dec;29(6):517-22. doi: 10.1016/s8756-3282(01)00614-7. PMID 11728921
- [Result] Bouxsein ML, Kaufman J, Tosi L, Cummings S, Lane J, Johnell O. Recommendations for optimal care of the fragility fracture patient to reduce the risk of future fracture. J Am Acad Orthop Surg. 2004 Nov-Dec;12(6):385-95. doi: 10.5435/00124635-200411000-00003. PMID 15615504
- [Result] Friedman SM, Mendelson DA. Fragility fractures. Clin Geriatr Med. 2014 May;30(2):xiii-xiv. doi: 10.1016/j.cger.2014.01.019. Epub 2014 Mar 4. No abstract available. PMID 24721376